CLINICAL TRIAL: NCT07342257
Title: A Randomized, Double-Blind, Active-Controlled, Phase I Clinical Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Zamerovimab and Mazorelvimab Injection (SYN023) in Combination With Rabies Vaccine in Healthy Subjects Under 18 Years of Age
Brief Title: SYN023 With Rabies Vaccine in Healthy Pediatric Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synermore Biologics (Suzhou) Co., Ltd. (Industry)
Collaborators: Guizhou Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYN023-007
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Rabies Post-exposure Prophylaxis
Keywords: rabies; pediatric; post-exposure prophylaxis; SYN023
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose SYN023 combined with rabies vaccine (Experimental): A single intramuscular injection of SYN023 at low dose combined with the Chinese licensed Vero Cell Rabies Vaccine (Essen 5-dose regimen)
  Interventions: Biological: SYN023; Biological: Rabies Vaccine
- High-dose SYN023 combined with rabies vaccine (Experimental): A single intramuscular injection of SYN023 at high dose combined with the Chinese licensed Vero Cell Rabies Vaccine (Essen 5-dose regimen)
  Interventions: Biological: SYN023; Biological: Rabies Vaccine
- HRIG combined with rabies vaccine (Active Comparator): A single intramuscular injection of Human rabies immunoglobulin (HRIG）combined with the Chinese licensed Vero Cell Rabies Vaccine (Essen 5-dose regimen)
  Interventions: Biological: Rabies Vaccine; Biological: HRIG

INTERVENTIONS:
Biological: SYN023 — SYN023 should be administered intramuscularly at sites distant from the vaccine injection site, either at the gluteus maximus or vastus lateralis muscles. The investigator should determine appropriate injection sites for multiple-point administration based on the participant's age and body weight. It is recommended that not more than 6 mL be administered per single gluteus maximus or vastus lateralis muscle, with not more than 4 mL per single injection site (younger children may require reduced volumes per muscle and per injection site based on individual circumstances); Injection time: Day 0.
  Other Names: Zamerovimab and Mazorelvimab Injection
  Arms: High-dose SYN023 combined with rabies vaccine; Low-dose SYN023 combined with rabies vaccine
Biological: Rabies Vaccine — Dosage and administration of Rabies vaccine for human use: 0.5 mL, intramuscular injection in the deltoid muscle; Injection time: Days 0, 3, 7, 14, and 28 (Essen 5-dose regimen).
  Other Names: Freeze-dried Rabies Vaccine for Human Use (Vero Cells)
Biological: HRIG — HRIG should be administered intramuscularly at sites distant from the vaccine injection site, either in the gluteus maximus or vastus lateralis muscles. The investigator should determine appropriate injection sites for multiple-point administration based on the participant's age and body weight. It is recommended that not more than 6 mL be administered per single gluteus maximus or vastus lateralis muscle, with not more than 4 mL per single injection site (younger children may require reduced volumes per muscle and per injection site based on individual circumstances); Injection time: Day 0.
  Other Names: Human Rabies Immunoglobulin
  Arms: HRIG combined with rabies vaccine

SUMMARY:
This study is a randomized, double-blind, active-controlled design. The goal is to evaluate the safety, pharmacokinetics and pharmacodynamic of SYN023 in combination with rabies vaccine in healthy participants under 18 years of age.

Participants will:

1. Be randomly assigned to receive one of two doses of SYN023 or a dose of HRIG by intramuscular injection on Day 0, along with the first dose of the rabies vaccine.
2. Receive additional doses of the rabies vaccine on Days 3, 7, 14, and 28.
3. Have all adverse events (within 42 days) and all serious adverse events (within 126 days) after PEP administration collected and recorded.
4. Provide several blood samples for pharmacokinetics and pharmacodynamic testing.

ELIGIBILITY:
Inclusion Criteria:

1. Under 18 years of age at enrollment, male or female, with legal identification available.
2. Legal guardians of the volunteers voluntarily agree to participate in the study and sign the Informed Consent Form (ICF). Specifically, for volunteers under 8 years old, ICF is signed by legal guardians while fully respecting the child's opinion; for volunteers aged 8-17 years, legal guardians sign the ICF while volunteers themselves sign the ICF for minor volunteers;
3. Willing and able to comply with all study procedures, expected to be able to complete all follow-up visits and maintain contact throughout the study period;
4. Female volunteers of childbearing potential must have a negative urine pregnancy test prior to investigational product/vaccine administration, be non-lactating, and agree to use effective contraception during the study;
5. In good general health with normal physical examination findings, vital signs measurements, and axillary temperature ≤ 37.0℃.

Exclusion Criteria:

1. Subjects with history of injection of rabies vaccine and/or rabies virus passive immunization agents such as equine immunoglobulin, equine purified F (ab') 2 fragment products and HRIG;
2. Subjects with history of being bitten by a dog, cat, ferret, fox, ferret, skunk, bat or raccoon (wound with skin damage) in the past 6 months;
3. Subjects who have had pyrexia (≥ 37.3℃) or other acute illness within 7 days before enrollment, or are in acute exacerbation of chronic diseases;
4. History or current presence of any autoimmune or immunodeficiency disorders (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid disease, HIV infection, etc.);
5. Subjects with loss of splenic function or functional impairment, such as asplenia due to any condition (e.g., splenectomy);
6. Subjects with a history of severe allergy to previous vaccination requiring medical intervention, such as generalized urticaria, allergic laryngeal edema, Henoch-Schonlein purpura, local allergic necrosis reaction (Arthus reaction), angioneurotic edema and anaphylactic shock; or known hypersensitivity to any component contained in the investigational products/vaccine;
7. History or current presence of any systemic disease or poorly controlled chronic condition that may interfere with safety or efficacy evaluations as determined by the investigator, including but not limited to hematologic disorders, hepatic/renal diseases, gastrointestinal disorders, respiratory diseases, malignancies, or history of major organ transplantation, etc.;
8. History or current presence of severe neurological disorders (e.g., epilepsy, convulsions or seizures [excluding febrile seizures], encephalopathy) or psychiatric illness, or family history of psychiatric disorders;
9. Presence of coagulation abnormalities (e.g., coagulation factor deficiency, platelet disorders);
10. Administration of immunoglobulins or blood products within 3 months prior to enrollment, or planned use during the study;
11. Receipt of systemic immunosuppressants or other immunomodulatory therapies within 3 months prior to enrollment, including but not limited to systemic corticosteroids (e.g., prednisone ≥ 2 mg/kg/day for > 2 weeks), or cytotoxic therapy, or planned administration during the trial;
12. Participation in other clinical trials within 3 months prior to enrollment, or planned participation during the study;
13. Administration of live-attenuated vaccines within 14 days or subunit/inactivated vaccines within 7 days prior to enrollment;
14. Presence of skin lesions, inflammation, ulcers, rashes, or scars at the intended injection site that may interfere with administration or local reaction assessment;
15. Any other condition considered by the investigator to render the participant unsuitable for study participation.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) and adverse events (AEs) | 42 days
Incidence of serious adverse events (SAEs) | 126 days

SECONDARY OUTCOMES:
Incidence of adverse reactions and adverse events | 30 minutes and 7 days
Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) | Days 3, 7, 14, 42, 98 and 126
  Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Percentage of Participants With Rabies Virus Neutralizing Activity (RVNA) ≥0.5 IU/mL | Days 3, 7, 14, 42, 98 and 126
  Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Area Under the Efficacy Curve for the Geometric Mean Concentration (GMC) of Rabies Virus Neutralizing Activity (RVNA) | Day 0 to Day 14
  Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT). Area Under the Efficacy Curve for the GMC of RVNA from Study Day 0 to Day 14 after administration (AUEC0-14)
Maximum serum concentration (Cmax) | 126 days
  Cmax for SYN023 mAb components CTB011 and CTB012 will be estimated at Day 0 (pre-dose), Day 3, Day 7, Day 14, Day 42, Day 98 and Day 126 post-dose, using non compartmental analysis.
Time to maximum concentration (Tmax) | 126 days
  Tmax for SYN023 mAb components CTB011 and CTB012 will be estimated at Day 0 (pre-dose), Day 3, Day 7, Day 14, Day 42, Day 98 and Day 126 post-dose, using non compartmental analysis.
Area under the concentration-time curve (AUC0-t and AUC0-∞) | 126 days
  AUC0-t and AUC0-∞ for SYN023 mAb components CTB011 and CTB012 will be estimated at Day 0 (pre-dose), Day 3, Day 7, Day 14, Day 42, Day 98 and Day 126 post-dose, using non compartmental analysis.
Terminal half-life (t1/2) | 126 days
  t1/2 for SYN023 mAb components CTB011 and CTB012 will be estimated at Day 0 (pre-dose), Day 3, Day 7, Day 14, Day 42, Day 98 and Day 126 post-dose, using non compartmental analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuping Dong Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou, China